CLINICAL TRIAL: NCT06948279
Title: Immediate Versus Elective Endoscopic Removal of Large Common Bile Duct Stones in High-Risk Elderly Patients
Brief Title: Immediate vs. Elective Endoscopic Removal of Large CBD Stones in High-Risk Elderly Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Liver Institute, Egypt (Other)
Responsible Party: Principal Investigator, Gasser Ibrahim El-Azab, Professor of Hepatology and Gastroenterology, National Liver Institute, Egypt
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 01066416087
Record Dates: First submitted 2025-04-21; First posted 2025-04-29 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-01

CONDITIONS: Choledocholithiasis; Jaundice, Obstructive
Keywords: Choledocholithiasis; Bile Duct; ERCP; Elderly
MeSH Terms: conditions — Choledocholithiasis; Jaundice, Obstructive | interventions — Cholangiopancreatography, Endoscopic Retrograde

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A (Stent-first Approach) (Active Comparator): Group A patients had a temporary plastic stent placed to facilitate bile drainage, with elective stone removal scheduled 8-12 weeks later.
  Interventions: Procedure: The endoscopic retrograde cholangiopancreatography (ERCP) with insertion of a plastic stent.
- Group B (Stone Retrieval-first Approach) (Placebo Comparator): In Group B, patients underwent immediate stone extraction attempts using conventional techniques such as basket, balloon, or mechanical lithotripsy as needed.
  Interventions: Procedure: The endoscopic retrograde cholangiopancreatography (ERCP) with immediate stone extraction attempts.

INTERVENTIONS:
Procedure: The endoscopic retrograde cholangiopancreatography (ERCP) with insertion of a plastic stent. — A plastic stent was placed during the initial ERCP, with elective stone removal scheduled 8-12 weeks later.
  Arms: Group A (Stent-first Approach)
Procedure: The endoscopic retrograde cholangiopancreatography (ERCP) with immediate stone extraction attempts. — Immediate ERCP for stone removal, utilizing conventional techniques such as basket, balloon, or mechanical lithotripsy as needed.
  Arms: Group B (Stone Retrieval-first Approach)

SUMMARY:
The goal of this clinical trial is to compare two different approaches for removing large or multiple stones from the common bile duct in older adults with chronic diseases. The main questions it aims to answer are:

Is it better to remove the stones immediately during the first endoscopic procedure? Or is it safer and more effective to place a temporary plastic stent first and remove the stones later?

Researchers will compare these two approaches to see which one leads to better stone clearance and fewer complications.

Participants will:

Undergo an endoscopic procedure (ERCP) to treat their bile duct stones. Be randomly assigned to either have immediate stone removal or have a stent placed first, with stone removal scheduled 8-12 weeks later.

Attend follow-up visits to monitor their recovery and check for complications.

This study is being conducted at the National Liver Institute, Menoufia University, Egypt.

DETAILED DESCRIPTION:
This study was designed to evaluate two different endoscopic treatment strategies for managing large or multiple common bile duct (CBD) stones in elderly patients considered high-risk due to age and comorbid conditions. The research was conducted at the National Liver Institute, Menoufia University in Egypt, a tertiary care center with a high volume of hepatobiliary cases and extensive expertise in endoscopic retrograde cholangiopancreatography (ERCP).

Study Design and Population This was a prospective, randomized, comparative clinical trial conducted between February 2022 and September 2024. A total of 400 patients aged 65 years or older, with a Charlson Comorbidity Index (CCI) ≥ 3 and radiologically confirmed large or multiple CBD stones, were enrolled. Large stones were defined as those with a diameter ≥15 mm; multiple stones were defined as three or more stones, each measuring ≥10 mm. Stone size and number were confirmed by computed tomography (CT) or magnetic resonance cholangiopancreatography (MRCP).

Eligible patients were randomly assigned in a 1:1 ratio to one of two groups:

Group A (Stent-first approach): Underwent initial biliary stenting followed by elective stone extraction 8-12 weeks later.

Group B (Stone retrieval-first approach): Underwent immediate endoscopic stone removal during the index ERCP.

Study Procedures and Intervention Details All participants underwent a standardized baseline assessment, including a comprehensive medical history, physical examination, laboratory testing (e.g., liver enzymes, complete blood count, coagulation profile), and imaging studies. Randomization was computer-generated and concealed from the enrolling clinical team to minimize selection bias. While blinding of patients and proceduralists was not feasible due to the nature of the interventions, outcome assessments-including imaging reviews and complication monitoring-were conducted by independent investigators who were blinded to treatment allocation.

ERCP procedures were performed using a side-viewing endoscope (Pentax ED-3490TK). In all patients, endoscopic sphincterotomy (EST) was performed, and selective CBD cannulation was achieved using standard or alternative techniques when necessary. In Group A, a 10 Fr, 10 cm plastic biliary stent was placed, with a follow-up ERCP scheduled after 8-12 weeks for elective stone removal. In Group B, stone extraction was attempted during the index ERCP using a balloon, Dormia basket, or mechanical lithotripsy. A stent was placed only if stone extraction was incomplete.

Calculation of Stone Burden CBD stone dimensions were measured from radiographic images, with adjustments for magnification using the endoscope diameter as a reference. The total stone burden, or stone index, was calculated as the sum of all stone diameters in centimeters. Two independent radiologists reviewed and averaged the measurements to ensure accuracy and objectivity.

Assessments and Follow-Up The primary outcome was the rate of complete stone clearance. Patients were monitored throughout hospitalization and followed at 2 weeks, 1 month, and 3 months after discharge. Follow-up evaluations included clinical examinations, laboratory testing (e.g., liver function, inflammatory markers), and repeat imaging studies. Complications were recorded in real time, and their severity was graded using established clinical criteria.

Statistical Analysis Plan The sample size was calculated to detect a 15% difference in stone clearance rates between the two groups, with 80% power and a two-sided alpha of 0.05. Statistical analysis was performed using SPSS software. Categorical variables were compared using the Chi-square test or Fisher's exact test, as appropriate. Continuous variables were assessed using Student's t-test or the Mann-Whitney U test, depending on the distribution. Statistical significance was defined as P < 0.05.

Ethical Considerations This study was approved by the Institutional Review Board of the National Liver Institute (Approval No. 00659) and conducted in accordance with the Declaration of Helsinki. Written informed consent was obtained from all participants or, when applicable, from their legal guardians.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 65 years
* Charlson Comorbidity Index (CCI) ≥ 3
* Presence of large or multiple CBD stones (defined as ≥1 stone ≥15 mm or ≥3 stones each ≥10 mm on imaging)
* Ability to provide informed consent (or via legal representative).

Exclusion Criteria:

* Contraindications to ERCP or general anesthesia
* History of biliary surgery or altered anatomy
* Benign or malignant strictures of the distal CBD
* Intrahepatic bile duct stones
* Moderate to severe cholangitis
* Malignancy or serious condition with life expectancy <6 months

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 400 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2024-09-01 (Actual)

PRIMARY OUTCOMES:
Rate of complete stone clearance | One month
  complete removal of all detectable stones from the common bile duct without the need for additional procedures

SECONDARY OUTCOMES:
ERCP-related adverse events | Three months
  The incidence of ERCP-related adverse events during hospitalization, the duration of the procedure, the length of hospital stay, the time from ERCP to discharge, the need for repeat ERCP procedures or alternative biliary interventions due to stone recurrence or complications, and the overall patient morbidity and mortality rates

CONTACTS AND LOCATIONS:
Overall Officials: Omkolsoum Alhaddad, M.D., Principal Investigator — National Liver Institute, Menoufia University Egypt.
Locations (1):
- National Liver Institute, Menoufia University, Egypt., Shebeen El-Kom, Monufia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No
There is no plan to share IPD for this study due to ethical and regulatory considerations, as well as the absence of a data-sharing infrastructure at our institution.

REFERENCES:
- [Background] Tonozuka R, Itoi T, Sofuni A, Itokawa F, Kurihara T, Tsuchiya T, Ishii K, Tsuji S, Ikeuchi N, Umeda J, Tanaka R, Honjyo M, Mukai S, Fujita M, Moriyasu F. Efficacy and safety of endoscopic papillary large balloon dilation for large bile duct stones in elderly patients. Dig Dis Sci. 2014 Sep;59(9):2299-307. doi: 10.1007/s10620-014-3156-9. Epub 2014 Apr 26. PMID 24771320
- [Background] Kim KH, Kim TN. Efficacy and Safety of Endoscopic Papillary Large Balloon Dilation for Removal of Large Bile Duct Stones in Advanced Age. Can J Gastroenterol Hepatol. 2016;2016:6568989. doi: 10.1155/2016/6568989. Epub 2016 Oct 12. PMID 27812520
- [Background] Ye X, Huai J, Sun X. Effectiveness and safety of biliary stenting in the management of difficult common bile duct stones in elderly patients. Turk J Gastroenterol. 2016 Jan;27(1):30-6. doi: 10.5152/tjg.2015.150305. Epub 2015 Dec 17. PMID 26674978
- [Background] Meng K, Zhang DY, Chen DX, Liu WJ, Fang KX, Chen S, Wu L, Li MY. Large common bile duct stones in high-risk elderly patients: Immediate endoscopic stone removal or elective stone removal? A single-center retrospective study. BMC Gastroenterol. 2023 Oct 5;23(1):344. doi: 10.1186/s12876-023-02976-0. PMID 37798726